CLINICAL TRIAL: NCT02118350
Title: Effect of Mat Pilates Training on Blood Pressure of Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Alessandra Medeiros, PhD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pilates
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mat Pilates training (Experimental): Mat Pilates training performed two times at week for 16 weeks.
  Interventions: Behavioral: Mat Pilates Training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mat Pilates Training — Mat Pilates training performed two times at week for 16 weeks.
  Arms: Mat Pilates training

SUMMARY:
The study aimed to evaluate the chronic effects of Mat Pilates Training on blood pressure, heart rate, double product and psychobiological factors in hypertensive medicated women and acute effects of Mat Pilates Exercise on blood pressure of such individuals.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensives women
* Age 30 to 59 years
* Nonactive
* Make use of antihypertensive medication

Exclusion Criteria:

* Orthopedic problems or other problem that prevented the exercises
* Change in drug treatment during protocol
* Absence in more than 25% of the exercise sessions

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 16 weeks
  Blood pressure was measured by Ambulatorial Monitoring Blood Pressure before and after trial period and by semiautomatic monitoring before and after a single session of Mat Pilates exercise.

SECONDARY OUTCOMES:
Heart Rate | 16 weeks
  Heart Rate was measured by Ambulatorial Monitoring Blood Pressure before and after trial period and by semiautomatic monitoring before and after a single session of Mat Pilates exercise.
Anxiety | 16 weeks.
  Anxiety was analyzed by State-Trait Anxiety Inventory (STAI), before and after trial period.
Stress | 16 weeks
  Stress was analysed by perceived stress questionnaire, before and after trial period.
Depression | 16 weeks
  Depression was analysed by Beck's Depression Inventory (BDI), before and after trial period.
Sleep quality | 16 weeks
  Sleep quality was analysed by The Pittsburgh Sleep Quality Index (PSQI), before and after trial period.
Perception of Sleep | 16 weeks
  Perception of Sleep was analysed by Mini Sleep Questionnaire, before and after trial period.
Sleepiness | 16 weeks
  Sleepiness was analysed by Epworth Sleepiness Scale, before and after trial period.
Quality of Life | 16 weeks
  Quality of Life was analysed by Questionnaire for Health-Related Quality of Life assessment of hypertensive patients, before and after trial period.
Flexibility | 16 weeks
  Flexibility was analysed by Bank of wells, before and after trial period.
Strength | 16 weeks
  Strength was analysed by hydraulic handgrip dynamometer, before and after trial period.
Body weight | 16 weeks
Height | 16 weeks
Waist circumference | 16 weeks
Hip circumference | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, Santos, São Paulo, Brazil